CLINICAL TRIAL: NCT02623712
Title: The Watch the Spot Trial: A Pragmatic Trial of More Versus Less Intensive Strategies for Active Surveillance of Patients With Small Pulmonary Nodules
Brief Title: The Watch the Spot Trial
Acronym: WTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); University of California, Davis (Other); University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Michael K Gould, MD, Professor, Kaiser Permanente
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 1000001
Record Dates: First submitted 2015-12-01; First posted 2015-12-08 (Estimated); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Solitary Pulmonary Nodule; Coin Lesion, Pulmonary; Lung Neoplasms; Carcinoma, Non-small-cell Lung
MeSH Terms: conditions — Solitary Pulmonary Nodule; Lung Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- More Frequent CT Surveillance (Active Comparator): Chest CT scans to be repeated at 3, 6, 12 and/or 24 months, depending on patient risk factors and nodule size and attenuation (density)
  Interventions: Other: More Frequent Surveillance Strategy
- Less Frequent CT Surveillance (Active Comparator): Chest CT scans to be repeated at 3, 6, 12 and/or 24 months, depending on patient risk factors and nodule size and attenuation (density). Overall, participants in the less frequent arm are expected to undergo 30% fewer surveillance imaging tests.
  Interventions: Other: Less Frequent Surveillance Strategy

INTERVENTIONS:
Other: More Frequent Surveillance Strategy — Chest CT scans to be repeated at 3, 6, 12 and/or 24 months, depending on patient risk factors and nodule size and attenuation (density)
  Arms: More Frequent CT Surveillance
Other: Less Frequent Surveillance Strategy — Chest CT scans to be repeated at 3, 6, 12 and/or 24 months, depending on patient risk factors and nodule size and attenuation (density). Overall, participants in the less frequent arm are expected to undergo 30% fewer surveillance imaging tests.
  Arms: Less Frequent CT Surveillance

SUMMARY:
This study will compare two clinically accepted protocols for surveillance imaging in individuals who are found to have a small pulmonary nodule on chest computed tomography (CT) scans.

DETAILED DESCRIPTION:
The investigators will conduct an unblinded, prospective, pragmatic, cluster-randomized, comparative effectiveness trial of more intensive versus less intensive CT surveillance of patients found to have small pulmonary nodules in diverse health care settings. The goal of this pragmatic clinical trial is to identify the surveillance strategy that will maximize early diagnosis for individuals with cancerous nodules, while minimizing unnecessary surveillance of patients without cancer that can result in emotional stress, exposure to harmful ionizing radiation, and the discovery of incidental findings that may lead to unnecessary treatment.

ELIGIBILITY:
Inclusion Criteria:

The target population includes adults with small lung nodules that may represent a new diagnosis of lung cancer, who typically would be managed by CT surveillance in usual clinical practice. Thus, we will enroll all patients:

* aged ≥35 years
* at least one nodule measuring ≤15 mm in average diameter on chest CT.

Exclusion Criteria:

* Pregnant Women
* Age <35 years
* Known diagnosis of cancer (except non-melanoma skin cancer) within 5 years

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34686 (Actual)
Dates: Start 2017-03-06 (Actual); Primary Completion 2024-09-04 (Actual); Study Completion 2024-09-04 (Actual)

PRIMARY OUTCOMES:
Proportion of cancerous nodules with tumor (T) stage greater than T1a disease by the AJCC staging system, 7th edition | 24 months after enrollment
  Among individuals with small pulmonary nodules identified either incidentally or by screening, compare more versus less intensive surveillance to determine the number of cancerous nodules that progress beyond T stage T1a.

SECONDARY OUTCOMES:
Number of days from date of nodule identification to date of cancer diagnosis | Up to 2 years
  Ongoing, final analysis in year 5
Survival time from date of cancer diagnosis until death or end of study | Up to 4 years
  Ongoing, final analysis in year 5
Emotional distress, measured with the Impact of Events Scale | Measured at 2 months, 13 months, and 25 months following nodule identification
  Compare patient-reported emotional distress
Anxiety, measured with the State Anxiety Inventory, 6-item | Measured at 2 months, 13 months, and 25 months following nodule identification
  Compare patient-reported anxiety
General health status, measured with a single question | Measured at 2 months, 13 months, and 25 months following nodule identification
  Compare patient-reported general health status
Numbers of imaging tests, biopsy tests and surgical procedures, measured by review of electronic health records | Measured from date of nodule identification until date of cancer diagnosis or completion of 24 months of follow-up
  Compare resource utilization.
Exposure to ionizing radiation, using the computed tomography dose index (CTDIvol), measured in mGy (milliGray) | Measured from date of nodule identification to date of cancer diagnosis or completion of 24 months of follow-up
  Compare effective radiation doses received.
Exposure to ionizing radiation, using the the dose length product (DLP), measured in mGy*cm | Measured from date of nodule identification to date of cancer diagnosis or completion of 24 months of follow-up
  Compare effective radiation doses received.
Numbers of CT scans recommended by the assigned protocol that were not ordered by the ordering provider, and/or not completed by the patient | Measured from date of nodule identification to date of cancer diagnosis or completion of 24 months of follow-up
  Compare adherence to the recommended protocols for CT surveillance, and adherence to use of low radiation dose techniques.

CONTACTS AND LOCATIONS:
Overall Officials: Michael K Gould, MD, MS, Principal Investigator — Kaiser Permanente School of Medicin
Locations (1):
- Kaiser Permanente Southern California, Pasadena, California, United States

IPD SHARING:
Plan to Share IPD: Yes
We plan to share de-identified IPD for all study variables with other researchers on request as long as there is an acceptable justification
Supporting Information: Study Protocol, SAP
Time Frame: De-identified IPD will be made available within 6-12 months following study completion, to allow time for the primary study team to complete manuscripts that report on each of the 4 study aims.
Access Criteria: Interested researchers will be required to submit a formal request with justification and aims to the study Data Coordinating Center. Requests will be reviewed and approved by the study Executive Committee. Relevant data use or data transfer agreements will need to be completed.

REFERENCES:
- [Background] MacMahon H, Austin JH, Gamsu G, Herold CJ, Jett JR, Naidich DP, Patz EF Jr, Swensen SJ; Fleischner Society. Guidelines for management of small pulmonary nodules detected on CT scans: a statement from the Fleischner Society. Radiology. 2005 Nov;237(2):395-400. doi: 10.1148/radiol.2372041887. PMID 16244247
- [Background] Naidich DP, Bankier AA, MacMahon H, Schaefer-Prokop CM, Pistolesi M, Goo JM, Macchiarini P, Crapo JD, Herold CJ, Austin JH, Travis WD. Recommendations for the management of subsolid pulmonary nodules detected at CT: a statement from the Fleischner Society. Radiology. 2013 Jan;266(1):304-17. doi: 10.1148/radiol.12120628. Epub 2012 Oct 15. PMID 23070270
- [Background] Gould MK, Donington J, Lynch WR, Mazzone PJ, Midthun DE, Naidich DP, Wiener RS. Evaluation of individuals with pulmonary nodules: when is it lung cancer? Diagnosis and management of lung cancer, 3rd ed: American College of Chest Physicians evidence-based clinical practice guidelines. Chest. 2013 May;143(5 Suppl):e93S-e120S. doi: 10.1378/chest.12-2351. PMID 23649456
- [Background] Berrington de Gonzalez A, Mahesh M, Kim KP, Bhargavan M, Lewis R, Mettler F, Land C. Projected cancer risks from computed tomographic scans performed in the United States in 2007. Arch Intern Med. 2009 Dec 14;169(22):2071-7. doi: 10.1001/archinternmed.2009.440. PMID 20008689
- [Background] Smith-Bindman R. Is computed tomography safe? N Engl J Med. 2010 Jul 1;363(1):1-4. doi: 10.1056/NEJMp1002530. Epub 2010 Jun 23. No abstract available. PMID 20573919
- [Background] Smith-Bindman R, Miglioretti DL, Johnson E, Lee C, Feigelson HS, Flynn M, Greenlee RT, Kruger RL, Hornbrook MC, Roblin D, Solberg LI, Vanneman N, Weinmann S, Williams AE. Use of diagnostic imaging studies and associated radiation exposure for patients enrolled in large integrated health care systems, 1996-2010. JAMA. 2012 Jun 13;307(22):2400-9. doi: 10.1001/jama.2012.5960. PMID 22692172
- [Background] Gould MK, Tang T, Liu IL, Lee J, Zheng C, Danforth KN, Kosco AE, Di Fiore JL, Suh DE. Recent Trends in the Identification of Incidental Pulmonary Nodules. Am J Respir Crit Care Med. 2015 Nov 15;192(10):1208-14. doi: 10.1164/rccm.201505-0990OC. PMID 26214244
- [Background] Wiener RS, Gould MK, Slatore CG, Fincke BG, Schwartz LM, Woloshin S. Resource use and guideline concordance in evaluation of pulmonary nodules for cancer: too much and too little care. JAMA Intern Med. 2014 Jun;174(6):871-80. doi: 10.1001/jamainternmed.2014.561. PMID 24710850
- [Background] Brenner DJ, Hall EJ. Computed tomography--an increasing source of radiation exposure. N Engl J Med. 2007 Nov 29;357(22):2277-84. doi: 10.1056/NEJMra072149. No abstract available. PMID 18046031
- [Background] Ost D, Fein AM, Feinsilver SH. Clinical practice. The solitary pulmonary nodule. N Engl J Med. 2003 Jun 19;348(25):2535-42. doi: 10.1056/NEJMcp012290. No abstract available. PMID 12815140
- [Derived] Gould MK, de Bie E, Qi L, Creekmur B, Mazzone PJ, Mularski RA, Ritzwoller DP, Slatore CG, Vachani A, Walter EC, Wiener RS, Dyer DS, McEvoy CE, Kelly K, Smith-Bindman R, Miglioretti DL; Watch the Spot Investigators. Baseline Characteristics of Participants and Pulmonary Nodules in the Watch the Spot Trial: A Pragmatic Trial of Less versus More Intensive Strategies for Active Surveillance of Patients With Small Pulmonary Nodules. Clin Lung Cancer. 2025 Sep;26(6):e472-e482.e1. doi: 10.1016/j.cllc.2025.05.011. Epub 2025 May 24. PMID 40518364
- [Derived] Gould MK, Creekmur B, Qi L, Golden SE, Kaplan CP, Walter E, Mularski RA, Vaszar LT, Fennig K, Steiner J, de Bie E, Musigdilok VV, Altman DA, Dyer DS, Kelly K, Miglioretti DL, Wiener RS, Slatore CG, Smith-Bindman R. Emotional Distress, Anxiety, and General Health Status in Patients With Newly Identified Small Pulmonary Nodules: Results From the Watch the Spot Trial. Chest. 2023 Dec;164(6):1560-1571. doi: 10.1016/j.chest.2023.06.022. Epub 2023 Jun 24. PMID 37356710

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-08-04): https://cdn.clinicaltrials.gov/large-docs/12/NCT02623712/Prot_SAP_002.pdf